CLINICAL TRIAL: NCT04604808
Title: Observational Prospective Study on the Effects of Hypoparathyroidism on Post-thyroidectomy Health-related Quality of Life (QoL-hPTP)
Brief Title: Study on the Effects of Hypoparathyroidism on Post-thyroidectomy Health-related Quality of Life (QoL-hPTP)
Acronym: QoL-hPTP
Status: Completed | Type: Observational
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Principal Investigator, Jose Luis Muñoz de Nova, Endocrine Surgeon Consultant, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Other Study IDs: QoL-hPTP
Record Dates: First submitted 2020-09-29; First posted 2020-10-27 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Hypoparathyroidism Postprocedural
Keywords: Health-related Quality of Life; Thyroidectomy; Postoperative hypoparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non hypocalcemic group: Patients that don't develop post-thyroidectomy hypocalcemia
- Hypocalcemic group: Patients that develop post-thyroidectomy hypocalcemia

SUMMARY:
Our study will evaluate the health related quality of life (HRQoL) after a thyroidectomy and the relevance of postoperative hypoparathyroidism. The patients submitted to a total thyroidectomy will be evaluated with three questionaries (SF-36, Hospital HADS and a specifically designed Likert-type questionary about the intensity of hypoparathyroidism symptoms). The first evaluation will be before the surgery, and the other two will be completed a week and a month after the procedure.

DETAILED DESCRIPTION:
Patients submitted to total thyroidectomy according to clinical practice will be invited to participate in this study. If they accept, they will have to complete three questionaries to evaluate their HRQoL: SF-36, Hospital Anxiety and Depression Scale (HADS) and a specifically designed Likert-type questionary about the intensity of hypoparathyroidism symptoms; the day before the surgery and one week and one month after it. In those cases that develop permanent hypoparathyroidism, an additional evaluation will be done 3, 6, 9 and 12 months after surgery.

Variables:

* Demographic variables: sex, age, BMI, personal background, previous treatment.
* Diagnosis variables: diagnosis, cytology (Bethesda System), preoperative laboratory values serum (albumin, glomerular filtrate rate, total and ionic calcium, phosphate, magnesium, parathormone (PTH), 25-hydroxide (OH) vitamin D, thyroid-stimulating hormone (TSH), T4, thyroid antibodies).
* Procedure variables: central compartment dissection, accidental parathyroidectomy, parathyroid autotransplant, surgery length, intraoperative complications.
* Post-operative variables:
* Laboratory test 24h after surgery: albumin, glomerular filtrate rate, total and ionic calcium, phosphate, magnesium, PTH, 25-OH vitamin D.
* Symptoms of Hypocalcemia: presence of spontaneous symptoms of hypocalcemia, such as paresthesias, and time from the surgery (measured in hours).
* Postoperative hypocalcemia: defined by a serum albumin-corrected calcium level below 8 mg/dL or by the presence of hypocalcemic symptoms that require calcium or vitamin D supplementation.
* Follow-up variables: all the patients will be evaluated one week and one month after surgery. When they develop a hypocalcemia, laboratory test will be repeated according to clinical practice. In all cases, this test will be repeated one month after surgery, together with thyroid function test. The need for oral supplementation of calcium and/or vitamin D analogs or even magnesium will be collected (doses and time needed). The definitive histological diagnosis and the number of additional parathyroid glands identified in the surgical specimen will be also collected. In cases that developed postoperative hypocalcemia, the investigators will record the time to resolution, defined as the absence of calcium or vitamin D supplementation and a PTH level above 13 pg/mL.

Statistical Analysis:

The patients will be divided into two group depending on the development of post-thyroidectomy hypoparathyroidism. The results of their HRQoL questionaries will be compared within both groups. The investigators will evaluate the influence of clinical variables on these results.

The quantitative variables that follow a normal distribution will be described by the mean and the standard deviation; and those who do not follow the normal distribution will be described by median and interquartile range. The qualitative variables will be defined by the number of events and the percentage. To know if the variable follow or not the normality the investigators will use de Kolmogorov-Smirnov test.

The quantitative variables with a normal distribution will be compared with Student t-test (if there are two means) or with ANOVA (for more than two means). To compare quantitative variables with a different distribution, the Mann-Whitney U test (2 means) or Kruskal-Wallis test (more than 2) will be use.

The association between quantitative variable with a normal distribution will be stablished by the Pearson correlation ratio; and for those who do not follow the normal distribution, with Spearman test.

χ2 test will be used to compare qualitative variables. If an absolute frequency less or equal to 5 is found in any of the contingency table cells, the Fisher's exact test will be used.

Every test will be considered if there is a minimum signification level of p<0,05.

Sample size calculation:

There is not enough published data in order to help us calculate a proper sample size. the investigators will conduce the first 40 patients as a pilot study, based on which it will estimate a definitive sample size. The investigators will take as reference the results of the SF-36 survey of the week after the surgery and a minimum difference to detect of the 10% of the punctuation.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to total thyroidectomy
* Patients older than 18 yo
* Patients who accept participating in the study.
* Patients who, before the surgery, have done a complete laboratory test.
* Patients followed for at least one month after surgery.

Exclusion Criteria:

- Patients submitted to a subtotal or completion thyroidectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients submitted to total thyroidectomy according to clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change in SF-36 score | Preoperative, one week and one month after surgery
  36-Item Short Form Health Survey questionnaire: 0 to 100 points, been a lower score a worse outcome
Change in HADS score | Preoperative, one week and one month after surgery
  Hospital Anxiety and Depression Scale: 0 to 42 points, been a higher score a worse outcome
Changes Questionary of hypocalcemia symptoms | Preoperative, one week and one month after surgery
  Specifical designed Liker-type questionary: Likert scale based score, from 1 to 10 points, been a higher score a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de La princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided